CLINICAL TRIAL: NCT02826252
Title: VENTASWITCH, Examination of Ventavis® (Iloprost) Inhalation Behavior Using the I-Neb® AAD® System in Patients With Pulmonary Arterial Hypertension When Switching the Iloprost Nebulizer Solution for Inhalation From 10 μg/mL (V10) to 20 μg/mL (V20)
Brief Title: Examination of Ventavis (Iloprost) Inhalation Behavior Using the I-Neb AAD System in Patients With Pulmonary Arterial Hypertension When Switching the Iloprost Nebulizer Solution for Inhalation From 10 μg/mL (V10) to 20 μg/mL (V20)
Acronym: VENTASWITCH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18838
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension (PAH)
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ventavis: The study will be conducted in patients who are enrolled in the German Ventavis patient support program Ventaplus.
  Interventions: Drug: Iloprost,(Ventavis, BAYQ6256); Device: I-Neb AAD system

INTERVENTIONS:
Drug: Iloprost,(Ventavis, BAYQ6256) — Ventavis (Iloprost) nebulizer solution for inhalation as 10 μg/mL (V10) and 20 μg/mL (V20).
Device: I-Neb AAD system — Nebulizer, allows digital recording of inhalation data such as doses, inhalations per day and duration of inhalation (per day) etc.

SUMMARY:
The aim of this study is to examine inhalation behavior in patients enrolled in the German Ventavis patient support program Ventaplus when these patients are switched from Ventavis (Iloprost) 10 μg/mL to Ventavis (Iloprost) 20 μg/mL formulation.

DETAILED DESCRIPTION:
The VENTASWITCH study will be a local, prospective and retrospective, observational, case-crossover study. Data are collected and downloaded from the I-Neb AAD (Adaptive Aerosol Delivery) System. Two data collection periods are planned: period one; data collection from the last 3 months using Ventavis (Iloprost) 10 μg/mL (V10) before the index date of switching to Ventavis (Iloprost) 20 μg/mL (V20) (retrospective part) and period two; data collection for 3 months using V20 from index date (prospective part).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years at time of signing informed consent.
* Patients, diagnosed with group 1 PAH.
* Patients must be enrolled in the German Ventavis patient support program Ventaplus.
* Patients who either already switched from V10 to V20 therapy or who agreed to do so according to their physician's decision.
* Patients must have been on V10 therapy for at least 2 weeks.
* Written informed consent must be obtained.

Exclusion Criteria:

- participation in other clinical or interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in patients who are enrolled in the German Ventavis patient support program Ventaplus which is executed for Bayer by the company Contra Care GmbH, Nürnberg. Patients who are enrolled in the program and repeatedly experienced extended inhalation times with Ventavis (Iloprost) 10 μg/mL which could possibly result in incomplete inhalations, are currently being switched to Ventavis (Iloprost) 20 μg/mL by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Number of inhalations on Iloprost 10 ug/mL and 20 ug/mL | Up to 6 months
Number of delivered doses (none/partial/full) on Iloprost 10 ug/mL and 20 ug/mL | Up to 6 months

SECONDARY OUTCOMES:
Inhalation durations (min) per session on Iloprost 10 ug/mL and 20 ug/mL | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany